CLINICAL TRIAL: NCT06011057
Title: Evaluation of Serum Levels of C Reactive Protein (CRP) and Its Correlation With Fetal Ultrasound Parameters in the Prediction of Threatened Miscarriage in the First Trimester
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, lecturer and consultant at Obstetrics and Gynecology Department., Al-Azhar University
Other Study IDs: Gyna._531
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Threatened Miscarriage
Keywords: threatened miscarriage; ultrasound parameters; C reactive protein; first trimester
MeSH Terms: conditions — Abortion, Threatened | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- threatened miscarriage Group: This group will include 50 pregnant women presenting with vaginal bleeding and/or abdominal cramps concerning for possible miscarriage in the first trimester. Inclusion criteria will be gestational age between 6-14 weeks by last menstrual period and/or ultrasound dating, and clinical signs/symptoms suggestive of threatened miscarriage including:
  Vaginal bleeding Abdominal cramps/pain Closed cervical os on exam Women with confirmed fetal demise on ultrasound will be excluded. Participants in this group will undergo blood testing to measure C reactive protein (CRP) level and fetal ultrasound to assess parameters like crown-rump length, heartbeat, yolk sac size, and embryonic motion. This group will provide data to assess C reactive protein (CRP) and ultrasound findings in women with threatened first trimester miscarriage.
  Interventions: Diagnostic Test: Serum C reactive protein (CRP) level; Diagnostic Test: Ultrasound
- Control Group: The control group will include 50 low-risk pregnant women matched to the threatened miscarriage group based on gestational age. Inclusion criteria are normal pregnancy dating, no vaginal bleeding/cramping, normal prior ultrasounds, and no history of pregnancy complications. Controls will undergo the same CRP blood testing and fetal ultrasounds as the threatened miscarriage group. This will provide comparative normal pregnancy CRP and ultrasound data. Matching controls on demographics and gestation will allow analysis of differences in CRP and ultrasound parameters between groups to determine predictors of pregnancy viability.
  Copy Retry
  Interventions: Diagnostic Test: Serum C reactive protein (CRP) level; Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Serum C reactive protein (CRP) level — An immunoturbidimetric method using a Modular P Analyzer will be used to carry out HSCRP assay, with a quantitation limit of 0.5 mg/L.
Diagnostic Test: Ultrasound — All examinations will be carried out by an experience operator with a transvaginal probe on high-resolution ultrasound machines. Pregnancies will be dated from the LMP. Other measurements will be obtained during the scan as the mean gestation sac diameter, volume of the gestation sac and the embryonic heart rate (FHR).

SUMMARY:
The goal of this observational study is to evaluate and compare in pregnant women with threatened miscarriage in the first trimester. The main questions it aims to answer are:

What is the correlation between serum C reactive protein (CRP) levels and fetal ultrasound parameters in predicting threatened miscarriage? How accurate are serum C reactive protein (CRP) levels versus ultrasound in predicting pregnancy loss in threatened miscarriage? Participants will have blood tests to measure C reactive protein (CRP) levels and fetal ultrasound exams to assess parameters like crown-rump length.

Researchers will compare serum C reactive protein (CRP) levels and fetal ultrasound findings to see if either or both can accurately predict pregnancy loss in women with first trimester threatened miscarriage.

DETAILED DESCRIPTION:
This observational study will enroll 100 pregnant women, with 50 in the threatened miscarriage group and 50 healthy controls, to compare serum C reactive protein (CRP) levels and fetal ultrasound findings for predicting early pregnancy loss.

Women presenting with first trimester bleeding and cramps concerning for threatened miscarriage will undergo blood testing to measure C reactive protein (CRP) levels and fetal ultrasound to assess parameters including crown-rump length, heartbeat, yolk sac size, and embryonic motion.

The control group will consist of 50 low-risk pregnant women without threatened miscarriage matched for gestational age. Controls will undergo the same blood and ultrasound assessments.

Researchers will compare serum C reactive protein (CRP) levels and ultrasound measurements between the threatened miscarriage and control groups. They will analyze which parameters differ significantly between groups and examine the predictive utility of C reactive protein (CRP) levels versus ultrasound for determining pregnancy viability.

Key outcomes will include correlation of C reactive protein (CRP) with ultrasound parameters, and diagnostic accuracy of C reactive protein (CRP) levels versus ultrasound in predicting pregnancy loss in threatened first trimester miscarriages.

This study aims to help optimize early pregnancy loss prediction and counseling for women with potential threatened miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women in the age group (20-35) between 7 and 13 weeks gestation in which a singleton embryo with evident cardiac activity with sure last menstrual period (LMP) constant with 1st trimester documented ultrasound
* The included subjects will be divided into two groups:-

  1. Group 1 (control) will consist of 50 pregnant women with uneventful pregnancies without any problem.
  2. Group 2 (patients) will consist of 50 pregnant women with threatened miscarriage, of them.

Exclusion Criteria:

* Multiple pregnancies.
* Women having received hormonal treatment or progesterone supplements.
* Pregnancies with a difference of more than 7 days between last menstrual period (LMP) and crown- rump length.
* History of general medical disease e.g. diabetes, thyroid disease or antiphospholipid syndrome, Presence of local (gynecological) disease e.g. fibroid or adnexal masses verified by normal appearance of the uterus and ovaries by ultrasound.
* Presence of uterine malformations e.g. hypoplastic uterus or septate uterus diagnosed by history of recurrent miscarriage, hysterosalpingography or 3D ultrasound, Intake of natural or synthetic progesterone.
* Obesity.
* Ectopic pregnancy
* Vesicular mole
* Fetal demise by Ultrasound

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study will only enroll pregnant women whose gender identity and biological sex assigned at birth are both female. Individuals who identify as any gender other than female will not be eligible, as the study is specifically assessing threatened miscarriage and pregnancy outcomes in women based on their biological sex. Eligible participants must self-identify and be biologically classified as female to align with the research questions on CRP levels, ultrasound findings, and pregnancy loss risk in women with threatened first trimester miscarriage.
Study Population: The study population will consist of 100 pregnant women, including 50 with threatened miscarriage and 50 healthy controls, recruited from obstetrics clinic at Al-Hussein University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Serum C reactive protein (CRP) levels in threatened miscarriage vs control groups | At enrollment (6-14 weeks gestation)
  Serum C-reactive protein (CRP) levels will be compared between the threatened miscarriage and control groups. CRP levels will be assessed from blood samples collected at the time of enrollment in the study (6-14 weeks gestation). The goal is to determine if CRP levels differ significantly between the threatened miscarriage and control groups and examine the correlation between C reactive protein (CRP) levels and threatened early pregnancy loss.

SECONDARY OUTCOMES:
Ongoing pregnancy | Ongoing pregnancy assessed at 24 weeks gestation
  Ongoing pregnancy rates at 24 weeks gestation will be compared between the threatened miscarriage and control groups.
miscarriage rates | pregnancy loss before 20 weeks
  Miscarriage rates, defined as pregnancy loss before 20 weeks, will also be compared between the two groups through completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Muhamed A Abdelmoaty, M.D., Principal Investigator — Al-Azhar University
Locations (1):
- Al-Hussein University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The sample size is small, so there is a risk of breaching participant privacy and identifiability even with de-identified data sets. We want to prioritize protecting patient confidentiality.
  Participants were not consented for broad data sharing, only for use of their data specifically for this study. Additional consent processes would be needed to enable sharing.
  There are logistical barriers around data de-identification, establishing a repository, and creating data use agreements which are beyond the scope of this study.
  The research questions can be adequately answered through analysis of aggregated data and publication of results. Sharing individual-level data is not necessary to achieve the specific aims.
  The sensitive nature of pregnancy loss data further underscores the need for confidentiality safeguards. Participants may not feel comfortable with their pregnancy information being shared widely.